CLINICAL TRIAL: NCT02952690
Title: Clinical Comparison of Different Stylet Angles for Orotracheal Intubation Using Glidescope® Video Laryngoscope in Children
Brief Title: Different Stylet Angles for Orotracheal Intubation Using Glidescope® Video Laryngoscope in Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Hee-Soo Kim, Professor, Seoul National University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: H1608-156-787
Record Dates: First submitted 2016-10-19; First posted 2016-11-02 (Estimated); Last update posted 2018-02-19 (Actual); Status verified 2018-02

CONDITIONS: Intubation

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- standard curve group (Active Comparator): The style is curved in accordance with the curve of GVL blade in this group.
  Interventions: Device: Glidescope® with standard-curved tip
- tip-manipulated curve group (Experimental): The style is curved in accordance with the curve of GVL blade and the distal tip of style is additionally bended to the left (15-20 degree) in this group.
  Interventions: Device: Glidescope® with tip manipulated stylet

INTERVENTIONS:
Device: Glidescope® with tip manipulated stylet — The intubating style is curved in accordance with the curve of GVL blade and the distal tip of style is additionally bended to the left (15-20 degree)
  Arms: tip-manipulated curve group
Device: Glidescope® with standard-curved tip — The style is curved in accordance with the curve of GVL blade
  Arms: standard curve group

SUMMARY:
The purpose of this study is to evaluate the feasibility of endotracheal intubation via glidescope videolaryngoscope (GVL) using different curve of stylet in 120 children aged between 1 and 5 year old.

DETAILED DESCRIPTION:
Pediatric patients aged 1-5 year old are randomly assigned to one of two groups; standard curve (S) and tip-manipulated curve (T) groups. After routine anesthetic induction, endotracheal intubation is performed with GVL. Size of GVL blade is selected according to weight; GVL 0: <1.5kg, GVL 1:1.5-3.6kg, GVL 2: 1.8-10kg, GVL 2.5: 10-28kg). Before intubation, stylet curve is differently manipulated according to group. The style is curved in accordance with the curve of GVL blade in S group, whereas the distal tip of style is additionally bended to the left (15-20 degree) in T group.

Time from visualization of glottis with GVL to approaching of endotracheal tube to glottis, and time to completion of intubation are measured. In addition, the easiness of intubation is assessed using Visual Analogue Scale (0: extremely easy, 10: extremely difficult) and will be compared in both groups.

ELIGIBILITY:
Inclusion Criteria:

1. children aged between 1 and 5 years who are scheduled for elective surgery
2. American Society of Anesthesiologist physical status I, II

Exclusion Criteria:

1. History of asthma
2. Active upper respiratory infection
3. Significant cardiopulmonary disease

Ages: 1 Year to 5 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 120 (Actual)
Dates: Start 2016-12 (Actual); Primary Completion 2017-04 (Actual); Study Completion 2017-04 (Actual)

PRIMARY OUTCOMES:
Time to tracheal intubation | up to 3 min after insertion of GVL
  From the insertion of GVL to completion of endotracheal intubation

SECONDARY OUTCOMES:
Time to approaching of endotracheal tube tip to glottis | up to 3 min after insertion of GVL
  From the insertion of GVL to approaching of endotracheal tube tip to glottis
Number of attempt for glottis passage of endotracheal tube | up to 3 min after insertion of GVL
The change in stylet angle | up to 3 min after insertion of GVL
  The number of additional manipulation of stylet for success of endotracheal intubation
Visual analogue scale for the easiness of endotracheal intubation | up to 3 min after insertion of GVL
  Measurement of the easiness of endotracheal intubation
Successful endotracheal intubation in 30 seconds | up to 3 min after insertion of GVL
  Success or failure in completion of endotracheal intubation in 30 seconds

CONTACTS AND LOCATIONS:
Locations (1):
- SNUH, Seoul, Jongro Gu, South Korea

IPD SHARING:
Plan to Share IPD: Undecided